CLINICAL TRIAL: NCT01962675
Title: Skilled Motor Training and tDCS to Improve Leg Function After Spinal Cord Injury
Acronym: SLT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left study institution, declined to continue study at new institution
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Edelle Field-Fote, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20110344
Record Dates: First submitted 2013-09-30; First posted 2013-10-14 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Spinal Cord Injury
Keywords: tDCS; motor training; SCI
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- tDCS and skilled training (Experimental): tDCS and skilled leg training. Transcranial direct current stimulation + step training TDCS will be delivered to the motor cortical area in conjunction with skilled locomotor training
  Interventions: Device: Transcranial direct current stimulation + step training; Behavioral: Sham transcranial direct current stimulation + step training
- Sham tDCS and skilled leg training (Sham Comparator): Sham (Non active) tDCS and skilled leg training. 'Sham transcranial direct current stimulation + step training Sham tDCS will be delivered to the motor cortical area in conjunction with skilled locomotor training
  Interventions: Behavioral: Sham transcranial direct current stimulation + step training

INTERVENTIONS:
Device: Transcranial direct current stimulation + step training — Direct current stimulation of motor cortex with low stimulation intensity
  Arms: tDCS and skilled training
Behavioral: Sham transcranial direct current stimulation + step training — Stepping over specified soft foam obstacles
  Other Names: Stepping training

SUMMARY:
The study investigates the effect of using transcranial direct current stimulation (tDCS) and skilled stepping training versus skilled stepping training with sham-tDCS in improving ankle and leg motor control in persons with ambulatory persons with spinal cord injury.

Hypotheses H1: Participants will display greater improvement in stepping function following tDCS combined with training compared to sham-tDCS and training.

H2: Participants will display greater gains in cortical excitability, as evidenced by lower cortico-motor threshold (MT) associated with the TA muscles following tDCS and training compared to following sham stimulation and training.

H3: Participants in the tDCS+training group will show greater increases walking speed in a timed 10 meter walking trial.

H4: Participants in the tDCS+training group will show be able to perform a greater number of toe-taps test.

DETAILED DESCRIPTION:
An estimated 265,000 individuals live with the consequences of SCI in the United States alone. Individuals with motor incomplete spinal cord injury (MISCI) commonly experience loss or impairment of lower extremity function. There are a limited number of options for restoration of walking function in individuals with motor-incomplete spinal cord injury (MISCI) who exhibit some ability to stand and walk but may be impeded by impaired voluntary control of the lower limb particularly, the ankle.

In persons with spinal cord injury, walking function is often limited by poor ability to lift and advance the legs. Lower extremity orthotic devices may be employed to stabilize the ankle joint and provide toe clearance during walking. However, these devices are cumbersome, and may be aesthetically unappealing.

Newer evidence indicates that non-invasive approaches to brain stimulation may provide a way to improve voluntary control of the legs and ankles in persons with neurologic disorders.

Purpose of this research study:

The overall goal of this study is to develop functional rehabilitation strategies that facilitate optimal restoration of leg and ankle motor control in individuals with MISCI. Individuals with MISCI exhibit some motor function below the level of lesion and include American Spinal Injury Association Impairment Scale (AIS) classifications AIS C and AIS D. We propose to test non-invasive cortical stimulation in combination with lower-extremity functional motor training for its ability to assist in improving fine motor control of the lower limbs in individuals with MISCI.

Studies have shown that non-invasive transcranial direct current stimulation (tDCS) can increase activity in specific cortical areas associated with motor learning, and therefore improve on the cortical and functional effects associated with motor practice training in individuals with SCI. If brain stimulation in combination with motor training is found to enhance improvements in control more effectively than motor training alone, this would provide a basis for further examining stimulation combined with lower limb joint therapy in individuals with spinal cord injury.

Objectives: To Assess improvements in lower extremity motor control that are associated with bilateral tDCS and functional motor training or sham tDCS and functional motor training in individuals with motor incomplete spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Motor incomplete Spinal cord injured subjects.
* Ability to walk 10 m with or without walking aides.
* Ability to Dorsiflex (Move foot up) at least 5 degrees from sitting.

Exclusion Criteria:

* Seizures
* Cognitive function impairment
* Brain surgery or intracranial metal implants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edelle C Field Fote, PhD, Principal Investigator — University of Miami
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew before assignment
Groups:
- Real tDCS - Sham tDCS: Real tDCS+skilled training
  Transcranial direct current stimulation + step training TDCS will be delivered to the motor cortical area in conjunction with skilled locomotor training
  Transcranial direct current stimulation + step training: Direct current stimulation of motor cortex with low stimulation intensity
  Step training: Stepping over specified soft foam obstacles
  Sham transcranial direct current stimulation + step training: Stepping over specified soft foam obstacles
  Sham tDCS+skilled training Sham (Non active) tDCS and skilled leg training. 'Sham transcranial direct current stimulation + step training Sham tDCS will be delivered to the motor cortical area in conjunction with skilled locomotor training
  Step training: Stepping over specified soft foam obstacles
- Sham tDCS - Real tDCS: Sham tDCS+skilled training
  Sham (Non active) tDCS and skilled leg training. 'Sham transcranial direct current stimulation + step training Sham tDCS will be delivered to the motor cortical area in conjunction with skilled locomotor training
  Step training: Stepping over specified soft foam obstacles
  Real tDCS+skilled training
  Transcranial direct current stimulation + step training TDCS will be delivered to the motor cortical area in conjunction with skilled locomotor training
  Transcranial direct current stimulation + step training: Direct current stimulation of motor cortex with low stimulation intensity
  Step training: Stepping over specified soft foam obstacles
Period: Overall Study
Arm/Group | Real tDCS - Sham tDCS | Sham tDCS - Real tDCS
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was to be PhD student dissertation. PI left institution. Months later PhD student withdrew without notice. Data were stored on computers and not accessible to PI. Computers were replaced by new lab director.
Groups:
- Total: Total of all reporting groups
Arm/Group | Real tDCS - Sham tDCS | Sham tDCS - Real tDCS | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Midswing Ankle ROM
Description: Measuring Ankle range of motion (ROM) first at Baseline and then up to 1 hour after intervention at the Midswing phase during Gait.
Time Frame: Two times, 1) Baseline, and 2) Up to 1 hour after intervention.
Population: as for baseline characteristics
Arm/Group | tDCS and Skilled Training | Sham tDCS and Skilled Leg Training
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change From Baseline Active Motor Threshold
Description: Measuring Active motor threshold using single pulse transcranial magnetic stimulation (TMS) of Motor cortex M1 area
Time Frame: Two times, 1) Baseline, and 2) Up to 1 hour after intervention.
Population: as for baseline characteristics
Arm/Group | tDCS and Skilled Training | Sham tDCS and Skilled Leg Training
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline Scores of a 10 m Walk Test
Description: Change from baseline score of the time required to perform 10 m walking.
Time Frame: Two times, 1) Baseline, and 2) Up to 1 hour after intervention.
Population: as for baseline characteristics
Arm/Group | Real tDCS - Sham tDCS | Sham tDCS - Real tDCS
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline Score on Toe Tap Test
Description: Measuring the Time required to perform toe taps
Time Frame: Two times, 1) Baseline, and 2) Up to 1 hour after intervention.
Population: as for baseline characteristics
Arm/Group | Real tDCS - Sham tDCS | Sham tDCS - Real tDCS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Study was to be PhD student dissertation. PI left institution. Months later PhD student withdrew without notice. Data were stored on computers and not accessible to PI. Computers were replaced by new lab director.
Arm/Group | tDCS and Skilled Training | Sham tDCS and Skilled Leg Training
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes